CLINICAL TRIAL: NCT03704935
Title: Long Term Effects and of a Pulmonary Rehabilitation Maintenance Program in Patients With a Chronic Respiratory Disease: Time Course and Determinants
Brief Title: Long Term Effects and of a Pulmonary Rehabilitation Maintenance Program
Acronym: LTAir+R
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0317
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Chronic Respiratory Disease
Keywords: Pulmonary rehabilitation; Maintenance program; Cohort; Microenvironment; Long-term benefits

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic respiratory diseases are characterized by a progressive and long term deline. Pulmonary rehabilitation (exercise training and therapeutic education) can improve several disease outcomes like dyspnea, exercise tolerance and health-related quality of life. After an inpatient PR program, maintenance program can stabilize the disease outcomes. However, maintenance program are heterogeneous and long term benefits (>36 month) have been observed in only one study, which is not feasible in France. A realistic maintenance program as proposed by the French Air+R network (http://airplusr.com/wordpress/) has only demonstrated benefits after 12 month. In addition, the time course of patients may be heterogeneous, with differens clusters that could be influenced by the clinical, functional and systemic determinants. In particular, the cellular muscle microenvironment could be deleterious for the muscle function in patients, caused by a "spill-over" of inflammatory pulmonary molecules in the systemic milieu.

ELIGIBILITY:
Inclusion criteria:

Patients with a chronic respiratory disease (COPD, Asthma, bronchiectasis , Fibrosis, Sleep Apnea, …) undergoing pulmonary rehabilitation (maintenance or inpatient)

Exclusion criteria:

Contraindication to exercise training

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a chronic respiratory disease (COPD, Asthma, bronchiectasis , Fibrosis, Sleep Apnea, …) undergoing pulmonary rehabilitation (maintenance or inpatient)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
6 minutes walking distance | 10 years
  6 minutes walking distance

SECONDARY OUTCOMES:
health-related quality of life | 10 years
  health-related quality of life : VQ-11 questionnaire
Forced expiratory volume in 1 seconde | 10 years
  Forced expiratory volume in 1 seconde : FEV1
BODE index | 10 years
  BODE index
death | 10 years
  death

CONTACTS AND LOCATIONS:
Overall Officials: Farés Gouzi, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Department of clinical Physiology - University Hospital, Montpellier, France